CLINICAL TRIAL: NCT03945565
Title: Effect of Intraoperative Oxygen Tension on Patient Outcomes After Off-pump Coronary Artery Bypass Grafting (the CARROT Trial)
Brief Title: FiO2 and Outcomes After OPCAB (the CARROT Trial)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Collaborators: Asan Medical Center (Other); Severance Hospital (Other)
Responsible Party: Principal Investigator, Yunseok Jeon, Professor of Anesthesiology and Pain Medicine, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: FiO2 OPCAB
Record Dates: First submitted 2019-04-08; First posted 2019-05-10 (Actual); Last update posted 2022-02-09 (Actual); Status verified 2022-02

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FiO2 0.3 (Active Comparator): Patients allocated to this group are going to receiving FiO2 of 0.3 during surgery
  Interventions: Other: Fraction of inspired oxygen level
- FiO2 0.8 (Active Comparator): Patients allocated to this group are going to receiving FiO2 of 0.8 during surgery
  Interventions: Other: Fraction of inspired oxygen level

INTERVENTIONS:
Other: Fraction of inspired oxygen level — A fraction of inspired oxygen level during off-pump coronary artery bypass grafting will be set differently between the study groups: 0.3 vs 0.8.

SUMMARY:
Conventionally, a relatively high level of fraction of inspired oxygen (FiO2) has been used for secure a margin of safety in patients undergoing cardiac surgery including off-pump coronary artery bypass grafting (OPCAB). Since the potential adverse effects of hyperoxemia (via reactive oxygen species, vasocontriction, perfusion heterogeneity, myocardiac injury, etc.), various studies on this topic has been performed. However, the results are conflicting and inconsistent, and the consensus about whether the use of additional oxygen supply in cardiac surgery has not been reached among practitioners yet. This study is a multicenter study (Seoul National University, Asan Medical Center, Severance Hospital) where the effect of different level of FiO2 on postoperative clinical outcomes is evaluated.

DETAILED DESCRIPTION:
A sub-study will also be conducted in part of patients of the present study. In 40 out of 500 (expected) patients, two different levels of FiO2 will be sequentially set with a 5-minute interval after the induction of general anesthesia. Mixed venous and regional cerebral oxygen saturation will then be recorded according to the change of FiO2.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for elective off-pump coronary artery bypass grafting

Exclusion Criteria:

* emergency
* robot-assisted surgery
* minimally invasive cardiac surgery requiring thoracotomy/one-lung anesthesia
* preoperative pulmonary morbidity requiring oxygen therapy
* preoperative use of ECMO or IABP
* preoperative tracheal intubation or mechanical ventilation

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 414 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2021-08-17 (Actual); Study Completion 2021-09-12 (Actual)

PRIMARY OUTCOMES:
hospital LOS | From the beginning of surgery until the hospital discharge after surgery through study completion, an expected average of two weeks
  length of hospital stay after off-pump coronary artery bypass grafting

CONTACTS AND LOCATIONS:
Overall Officials: Yunseok Jeon, Principal Investigator — Seoul National University Hospital
Locations (1):
- Department of Anesthesiology and Pain Medicine, Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Nam K, Nam JS, Kim HB, Chung J, Hwang IE, Ju JW, Bae J, Lee S, Cho YJ, Shim JK, Kwak YL, Chin JH, Choi IC; CARdiac suRgery and Oxygen Therapy (CARROT) Investigators; Lee EH, Jeon Y. Effects of intraoperative inspired oxygen fraction (FiO2 0.3 vs 0.8) on patients undergoing off-pump coronary artery bypass grafting: the CARROT multicenter, cluster-randomized trial. Crit Care. 2023 Jul 13;27(1):286. doi: 10.1186/s13054-023-04558-8. PMID 37443130